CLINICAL TRIAL: NCT00656721
Title: Flutter Valve Improves Respiratory Mechanics and Sputum Production in Bronchiectasis Patients
Brief Title: Respiratory Mechanics Effects of Flutter Valve in Bronchiectasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Fernando Silva Guimaraes, Associate Professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 002434-UFRJ
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; physiotherapy; flutter valve; impulse oscillation technique
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flutter Valve (Experimental): This a crossover study, so all subjects performed both, control and experimental interventions. In Flutter Valve intervention the subjects remained comfortably seated, breathing through the device for 15 minutes, starting off from the total pulmonary capacity, and being free to cough. Thereafter, a 5-min session of cough ensued. In the control intervention the subjects followed the same sequence of the Flutter Valve intervention, but the metallic sphere and the cover of the device were removed. Since the patients were not acquainted with the valve, they did not know its proper assembly. As in the Flutter Valve intervention, during 15 minutes the patients could expectorate spontaneously and return to the device. A 5-min coughing session took place.
  Interventions: Device: Flutter Valve

INTERVENTIONS:
Device: Flutter Valve — Flutter Valve (Scandipharm, Birmingham, AL) is shaped like a pipe with a hardened plastic mouthpiece at one end, a plastic protective, perforated cover at the other end, and a high-density stainless steel ball resting in a plastic circular cone on the inside. When the patient expires, a vibratory effect is transmitted to airways by the steel ball oscillation in order to facilitate mucociliary clearance.
  In our study, the use of the equipment was guided by a registered physical therapist, but the position (angle) was determined by the patient, according to his/her adaptation and perception of effectiveness of sputum clearance. The patients remained comfortably seated, breathing through the device for 15 minutes, starting from the total pulmonary capacity, and being free to cough. Thereafter, a 5-minute session of cough was done.
  Other Names: FLUTTER® Mucus Clearance Device

SUMMARY:
Considering that respiratory physiotherapy lack scientific evidence to support its application in the treatment of several obstructive diseases, this investigation was designed to evaluate the hypothesis that Flutter Valve can improve the airway clearance of hypersecretive bronchiectasis patients.

DETAILED DESCRIPTION:
The application of airway clearance techniques is considered an important component in the treatment of bronchiectasis patients (Van der Shans, 1997). For this purpose, a number of techniques has been introduced in the last decades. The Flutter Valve was initially proposed for the treatment of children with cystic fibrosis (CF) (Lindemann, 1992), but there is not enough evidence about its utilization in patients with bronchiectasis (Van der Shans & cols, 1999).

The effects of the Flutter Valve on respiratory mechanics of patients with bronchiectasis have been evaluated by forced spirometry (Pryor e cols, 1994; Gondor e cols, 1999; Thompson e cols, 2002). This approach however, does not allow the characterization of mucus transportation along the airways (Williams, 1994). The forced oscillation technique (FOT), a non-invasive alternative to characterize respiratory mechanics, allows the evaluation of respiratory mechanics at different frequencies without special maneuvers (Dubois e cols., 1956). According to eligibility criteria and in a randomized order, the patients were submitted to two protocols (control and Flutter Valve intervention), with one-week interval between them (washout). Respiratory mechanics and expectorated sputum volume were assessed before and after each intervention, in order to assess the Flutter Valve effect on tracheobronchial sputum removal.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical and high-resolution computerized tomography diagnosis.

Exclusion Criteria:

* chest pain,
* acute hemoptysis,
* recent history of rib fracture or pneumothorax (less than 1 year),
* respiratory infection in the four weeks before measurements,
* asthma,
* cystic fibrosis,
* daily sputum production lower than 25 mL/day

Ages: 28 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Expectorated sputum volume. | After each evaluated procedure (control and Flutter Valve intervention)

SECONDARY OUTCOMES:
Respiratory mechanics (spectral data recorded by impulse oscillation technique). | Before and after each applied procedure (control and Flutter Valve intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando S Guimarães, PhD, Study Chair — Universidade Federal do Rio de Janeiro
Locations (2):
- Brazil (2):
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro